CLINICAL TRIAL: NCT01806662
Title: Randomized Pilot Study of Ustekinumab for Subjects With Chronic Atopic Dermatitis Who Have Sub-optimal Response to Prior Therapy
Brief Title: Pilot Study of Ustekinumab for Subjects With Chronic Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: JKR-0737
Record Dates: First submitted 2013-02-28; First posted 2013-03-07 (Estimated); Results first posted 2017-12-19 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-02

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Arm (Ustekinumab first, Then Placebo) (Experimental): Since there is a crossover design, each patient will be in the treatment arm for 16 weeks of the study.
  Interventions: Drug: Ustekinumab; Other: Placebo
- Placebo Arm (Placebo first, Then Ustekinumab) (Placebo Comparator): Since there is a crossover design, each patient will be in the placebo arm for 16 weeks of the study. If a patient begins in the placebo arm, they will switch over to the treatment arm at week 16.
  Interventions: Drug: Ustekinumab; Other: Placebo

INTERVENTIONS:
Drug: Ustekinumab — Injection of monoclonal antibody against the p40 subunit of IL-12/23
  Other Names: Stelara
Other: Placebo — Injection of placebo

SUMMARY:
Atopic dermatitis (AD) is a chronic disease associated with intense itching, which affects most aspects of everyday life in the majority of patients. Acute inflammation and extensor/facial involvement is common in infants, whereas chronic inflammation increases in prevalence with age, as do localization to flexures. AD has a complex background characterized by immune activation, increased epidermal thickness in chronic diseased skin, and defective barrier function. In normal, healthy skin, the outer layer of the epidermis, the stratum corneum is made up flattened dead cells called corneocytes held together by a mixture of lipids and proteins. The stratum corneum and, in particular, the lipid layer are vital in providing a natural barrier function that locks water inside the skin and keeps allergens and irritants out. In people with AD, the barrier function is defective, which leads to dry skin. As the skin dries out, it cracks allowing allergens and irritants to penetrate.

Mild AD can be controlled with emollients and topical medications. However, moderate to severe AD is extremely difficult to control and requires systemic treatment that is often unsatisfactory due to impracticality and lack of effectiveness. Only three therapeutic options exist for moderate to severe AD, including: 1) oral steroids 2) cyclosporine A (CsA), that is not widely used in the US as it is not FDA approved for AD and 3) ultraviolet phototherapy. Oral steroids and CsA treatments have major side effects and UV radiation therapy is highly inconvenient for patients. Several biologic medications, such as TNF-alpha inhibitors, are effective, convenient, and relatively safe therapies for psoriasis, but have thus far not shown efficacy in AD. Ustekinumab is a unique biologic medication that may specifically target AD.

The investigators study will determine whether there is a reversal of the skin thickness and the immune pathways involved in the disease during treatment with Ustekinumab and what specific immune cells are involved. The investigators are also interested to understand how the clinical reversal of the disease will correlate with tissue reversal of the disease.

DETAILED DESCRIPTION:
In psoriasis, epidermal hyperplasia is driven by underlying immune activation, whether as a direct response to IL-20 family cytokines that induces hyperplasia and inhibits keratinocyte terminal differentiation or as an indirect response to immune-mediated injury to keratinocytes. The epidermal reaction in psoriasis is largely restored to normal with selective immune suppression. Hence, one might hypothesize that similar epidermal responses should occur in the presence of "generalized" cellular immune activation, in diseases with similar inflammatory infiltrate and epidermal hyperplasia, such as AD. In fact, psoriasis and AD share features of dense T-cells and dendritic cell infiltrates, as well as over-expression of IL-22 in skin lesions. These diseases also share similar epidermal hyperplasia in their chronic phases.

Work from the investigators group showed that IL-22 is a key cytokine in the pathogenesis of both AD and psoriasis. The investigators have demonstrated that in psoriasis, ustekinumab suppresses the production of IL-12, IL-23, and IL-22. Additionally, by RT-PCR the investigators demonstrated that the mRNA expression of p40 cytokine and the IL23R is up-regulated in AD as compared to both normal skin and psoriasis. The investigators therefore hypothesize that ustekinumab will suppress IL-22 and possibly also p40 production in AD lesions and reverse both the epidermal growth/differentiation defects and the underlying immune activation, and hence will suppress disease activity. Interestingly, p40 was also found to be significantly up-regulated in non-lesional AD skin as compared with normal skin.

Although AD is thought to be predominately a disease of Th2-type cells, in the chronic stage, there is large Th1 component. To date, the precise mechanism by which sequential activation of Th2 and Th1 cells in AD is achieved remains unknown. IL-12 induces the differentiation and maturation of human Th cells into Th1-type cells. Recent circumstantial evidence suggests that in AD patients IL-12 may facilitate a change from the Th2-type to a Th1 cytokine profile. IL-12 was recently shown to be highly elevated in pediatric AD and its levels were strongly associated with disease severity.

Expression of IL-12 p40 mRNA is significantly enhanced in lesional skin from AD, suggesting that the enhanced local production of IL-12 in dendritic cells and macrophages may be responsible for the increased production of IFN-γ in chronic lesions potentially suggesting that IL-12 may have a pivotal role in promoting inflammation in atopic dermatitis. Topical steroids which constitute a mainstay of therapy in AD are known to strongly down-regulate IL-12 expression, possibly also indicating that targeted anti IL-12 therapy might important role in treating AD.

Recently, the Th1/Th2 paradigm in autoimmunity and allergy has been revisited to include a role for a new population of IL-17-producing Th cells known as Th17. Th17 cells are characterized by the production of inflammatory cytokines such as IL-17A, IL-17F, IL-22, and IL-26. One of the key factors involved in naive Th-cell commitment to a Th17 phenotype is IL-23.

Patients with acute AD were found to have increased Th17 T-cells in peripheral blood by flow cytometry and intracellular cytokine staining 26 as well as by immunohistochemistry (IHC) in lesions. Since IL-23 is the major inducer of Th17 T-cells, as well as "T22" T-cells, neutralization of IL-23 could potentially result in both decreased Th17 signal in acute AD as well as decreased "T22/IL22" signal. Therefore the investigators postulate that ustekinumab in AD will act both inhibiting the IL-12-dependent Th1 shift in chronic AD stage as well as the pathogenic IL-22/"T22" axis in this disease.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female and ages 18-75.
* Have moderate to severe AD (as determined using the Objective SCORAD scale ≥15) and a history of therapeutic failure with at least two of the three different treatment categories as listed within the inclusion criteria.
* Patients must have tried and failed at least two of the three treatment categories of the following treatment modalities:

Category 1 : Hydration plus topical steroids and/or antibiotics Category 2: Systemic Steroids and/or Phototherapy Category 3: Cyclosporine and/or Other Immunomodulators (Methotrexate, CellCept, Immuran, topical Calcineurin inhibitors)

* Patients who initially respond to cyclosporine but cannot sustain a response after the drug is discontinued will also be eligible.
* Patients that have contraindications to category 3 drugs will also be allowed to participate in the study.
* A washout period prior to screening will be required for the following medications:
* Cyclosporine/Oral Steroids/Imuran/Mycophenolate Mofetil/Other systemic immunosuppressants: 4 weeks
* Phototherapy/Moderate to High Potency Topical Corticosteroids: 2 weeks
* Women of childbearing potential must test negative for pregnancy and be using adequate birth control measures (e.g., Abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, or have had a tubal ligation or a hysterectomy) during the study and for 6 months after receiving the last treatment. Likewise, men capable of fathering children must also use appropriate methods of birth control (e.g., abstinence, barrier methods with spermicide, or have had surgical sterilization such as vasectomy).
* Patients must be in general good health in the opinion of the investigator.
* Patients with stable chronic asthma, treated with inhaled corticosteroids, will be eligible.
* The screening laboratory tests must meet the following criteria:

Hemoglobin >9 g/dl WBC count >3.5 x 109 cells/L Neutrophils >1.5 x 109 cells/L Platelets >100 x 109 cells/L AST/SGOT and ALT/SGPT levels must be within 2 times the upper limit of normal for the laboratory conducting the test. Alkaline phosphatase levels must be within 2 times the upper limit of normal for the laboratory conducting the test.

* Are PPD negative at the time of screening.
* The patients will be allowed to use topical therapy during the washout period. These will include emollients, and mild steroids (class 6 or 7), except on one target area that will be the site for the skin biopsies.

Exclusion Criteria:

* Previous treatment with ustekinumab or other agent that specifically targets IL-12 or 23
* Have a history of latent or active granulomatous infection, including TB, histoplasmosis, or coccidioidomycosis, prior to screening, or are frequently in contact with individuals who carry active TB infection or a non-tubercular mycobacterial infection or an opportunistic infection
* Are HIV positive by history or POCT on the screening visit
* Have documented current active hepatitis B (surface antigen positive or asymptomatic chronic carriers) or hepatitis C infection (anti-HCV positive), by history and/or screening test
* Have a history of substance abuse (drug or alcohol) within the past year before screening
* Have any serious concomitant illness that could require the use of systemic corticosteroids or otherwise interfere with the patient's participation in the trial
* Pregnant women or women that are breast-feeding or plan to breast feed. Women of childbearing age who plan to get pregnant within 15 weeks of stopping study agent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Krueger, MD PhD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm (Ustekinumab First, Then Palcebo): Since there is a crossover design, each patient will be in the treatment arm for 32 weeks (16 weeks on Ustekinumab, then 16 weeks on Placebo) of the study.
  Ustekinumab: Injection of monoclonal antibody against the p40 subunit of IL-12/23
- Placebo Arm (Placebo First, Then Ustekinumab): Since there is a crossover design, each patient will be in the placebo arm for 16 weeks of the study. If a patient begins in the placebo arm, they will switch over to the treatment arm at week 16 (for 16 weeks).
  Placebo: Injection of placebo
Period: First Intervention (Weeks 0-16)
Arm/Group | Treatment Arm (Ustekinumab First, Then Palcebo) | Placebo Arm (Placebo First, Then Ustekinumab)
Started | 16 | 16
Received Intervention | 12 | 15
Completed | 12 | 15
Not Completed | 4 | 1
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Adverse Event | 0 | 1
Period: Second Intervention (Weeks 16-32)
Arm/Group | Treatment Arm (Ustekinumab First, Then Palcebo) | Placebo Arm (Placebo First, Then Ustekinumab)
Started | 12 | 15
Completed | 10 | 11
Not Completed | 2 | 4
Not completed — Lack of Efficacy | 2 | 3
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Since there is a crossover design, each participant will be in the Treatment Arm (Ustekinumab first, Then Placebo) or Placebo Arm (Placebo first, Then Ustekinumab) for 16 weeks of the study. They will crossover to the other treatment at week 16 for 16 weeks (32 weeks total).
  Placebo: Injection of placebo Ustekinumab: Injection of monoclonal antibody against the p40 subunit of IL-12/23
Arm/Group | All Study Participants
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 38.5 [18 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of SCORAD-50 Response at Week 16.
Description: Greater improvement from their baseline objective SCORAD (SCORing Atopic Dermatitis) at Week 16. The efficacy variable for each randomized group is the proportion of subjects who achieve an improvement of 50% or greater from their baseline objective SCORAD at Week 16 (at crossover). SCORAD-50 is the percentage of decrease in baseline SCOARD at Week 16.
  SCORAD is a clinical tool used to assess the extent and severity of eczema. Calculation is based on extent of involvement (skin involvement) and subjective symptoms of itching and loss of sleep. The SCORAD scale ranges from 0 (minimum, lowest possible score, Mild severity) to 103 (maximum, highest possible score, Severe severity) [last observation carry forward].
Time Frame: Week 16
Population: Proportion of participants with improved outcome.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Arm (Ustekinumab First, Then Palcebo): Since there is a crossover design, each patient will be in the treatment arm for 16 weeks of the study.
  Ustekinumab: Injection of monoclonal antibody against the p40 subunit of IL-12/23
Arm/Group | Treatment Arm (Ustekinumab First, Then Palcebo) | Placebo Arm (Placebo First, Then Ustekinumab)
Number analyzed (Participants) | 16 | 16
Participants | 5 | 3

ADVERSE EVENTS:
Time Frame: 16 weeks for each intervention.
Description: Adverse Event reporting included all participants who received at least one dose of intervention.
Groups:
- Ustekinumab: Participants who received Ustekinumab injection for 16 weeks.
  Ustekinumab: Injection of monoclonal antibody against the p40 subunit of IL-12/23
- Placebo: Participants who received Placebo injection for 16 weeks.
  Placebo: Injection of placebo
Arm/Group | Ustekinumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 4/32 | 10/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ustekinumab (N=32) | Placebo (N=32)
upper respiratory infection (General disorders) | 3 (3) | 1 (1)
ear infection (Ear and labyrinth disorders) | 1 (1) | 0 (0)
fall (General disorders) | 1 (1) | 1 (1)
musculoskeletal pain (General disorders) | 1 (1) | 1 (1)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Contact dermatitis/allergy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema herpeticum flare (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Light Headed (Nervous system disorders) | 1 (1) | 0 (0) — Lightheadedness after biopsy
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) — Infection: other: Pulmonary/Respiratory: Lungs
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) — Infection: Other: Renal/Genitourinary: Urinary Tract
Eczema Flare (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Diaphoresis (Immune system disorders) | 0 (0) | 1 (1) — Allergy/Immunology
Blood per rectum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flu-like symptoms (General disorders) | 0 (0) | 1 (1) — Flu-like Syndrome
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) — Pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No